CLINICAL TRIAL: NCT03466112
Title: Aerobic Exercise for the Improvement of Cognition and Enhancement of Recovery in Post-acute Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: RWTH Aachen University (Other); Charite University, Berlin, Germany (Other); Heinrich-Heine University, Duesseldorf (Other); Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Principal Investigator, Prof. Peter Falkai, Prof. Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Version (V) 2.0 - 30.07.2018
Record Dates: First submitted 2018-02-19; First posted 2018-03-15 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
Keywords: exercise
MeSH Terms: conditions — Schizophrenia; Motor Activity | interventions — Endurance Training; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- endurance training (Experimental): endurance training with stationary bicycles
  Interventions: Other: endurance training
- balance and tone program (Active Comparator): flexibility, core strength, balance, relaxation
  Interventions: Other: balance and tone program

INTERVENTIONS:
Other: endurance training — endurance training with stationary bicycles
  Other Names: aerobic exercise
  Arms: endurance training
Other: balance and tone program — flexibility, core strength, balance, relaxation
  Arms: balance and tone program

SUMMARY:
The study investigates the efficacy of aerobic exercise on cognitive performance and brain plasticity in schizophrenia.

DETAILED DESCRIPTION:
This multi-center, two-arm, parallel-group, randomized placebo-controlled add-on clinical trial investigates the efficacy of aerobic exercise on cognitive performance and brain plasticity in schizophrenia. The aim is the enhancement of recovery with the use of 26 weeks of continuos endurance training (aerobic exercise) with stationary bicycles or a balance and tone program consisting of exercises for flexibility, core strength, balance and relaxation. Followed by a follow-up period of 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given by the subject; DSM-IV-TR diagnosis of schizophrenic psychosis (295.10-30, 295.90); age 18 to 65 years, male or female; PANSS at baseline: total score ≤ 75, proper contraception in female patients of childbearing potential; treatment with one or two antipsychotics in a stable dose of at least two weeks, body mass index between 18 and 40.

Exclusion Criteria:

* Lack of accountability; positive urine drug-screening for illicit drugs at screening (except benzodiazepines); serious suicidal risk at screening visit; other relevant interferences of axis 1 according to diagnostic evaluation (MINI); other relevant neurological or other medical disorders; pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
all-cause discontinuation | 12 months (at baseline, day 14, 68, 98, 140, 182, 196, 273 and day 365)
  Reason of study discontinuation will be identified. The all-cause-discontinuation questionnaire will be called up 9 times from baseline up to 12 months (compare time frame) including 26 weeks of intervention and 26 weeks follow up period. Reasons are defined as (1) relevant worsening of clinical symptoms (PANSS total score above 75 on cancerous visits for more than 14 days. (2) failure to take the prescribed medication for more than 14 days. (3) Failure to comply scheduled study or diagnostic appointments for more than 6 weeks (4) Patient unavailability despite extensive efforts of the treatment team (5) Withdrawal of patient consent (6) Clinician discontinuation.

SECONDARY OUTCOMES:
improvement in neurocognition (VLMT) | 12 months (at baseline, day 98, day 182 and day 365)
  As part of the measurement of cognitive performance during the screening phase and at the main measurement times (at baseline, day 98, day 182 and day 365), patients and control subjects will be tested using the Verbal Learning and Memory Test (VLMT).
improvement in neurocognition (DSST) | 12 months (at baseline, day 98, day 182 and day 365)
  As part of the measurement of cognitive performance during the screening phase and at the main measurement times (at baseline, day 98, day 182 and day 365), patients and control subjects will be tested using a test of verbal declarative episodic memory, the Digit Symbol Substitution Test (DSST).
improvement in neurocognition (TMT) | 12 months (at baseline, day 98, day 182 and day 365)
  As part of the measurement of cognitive performance during the screening phase and at the main measurement times (at baseline, day 98, day 182 and day 365), patients and control subjects will be tested using the Trail Making Test A and B (TMT) as a test of executive functions, quick visual comprehension, attention, and processing speed.
improvement in neurocognition (B-CATS) | 12 months (at baseline, day 98, day 182 and day 365)
  The partial aspect of verbal fluid from the letter Cognitive Assessment Tool for Schizophrenia (B-CATS) is also used in the neuropsychological investigation at the main measurement times (at baseline, day 98, day 182 and day 365).
improvement in neurocognition (MASC) | 12 months (at baseline, day 98, day 182 and day 365)
  As part of the measurement of cognitive performance during the screening phase and at the main measurement times (at baseline, day 98, day 182 and day 365), patients and control subjects will be tested using the Facial Affect Recognition (AOP) and Theory of Mind methods. These are tasks using the Movie for the Assessment of Social Cognition (MASC).
improvement in psychopathology (PANSS) | 12 months (At baseline, day 98, 182 and day 365)
  The assessment of psychopathology on the basis of a patient interview takes place at all main measurement times. At baseline, day 98, 182 and day 365. The PANSS uses a standard procedure for assessing schizophrenia symptoms, which measures the severity of individual symptoms as well as the various symptom subgroups of positive and negative symptoms and general psychopathology.
improvement in psychopathology (CGI) | 12 months (at baseline, day 14, 68, 98, 140, 182, 196, 273 and day 365)
  The Clinical Global Impression Scale (CGI) assesses the overall symptom severity and response to interventions or therapies for psychiatric conditions to assess the effectiveness of the measures applied. It will be called up 9 times from baseline up to 12 months: At baseline, day 14, 68, 98, 140, 182, 196, 273 and day 365.
improvement in psychopathology (SOFAS) | 12 months (at baseline, day 14, 68, 98, 140, 182, 196, 273 and day 365)
  The Social and Occupational Functioning Assessment Scale (SOFAS) estimates social and professional performance. It will be called up 9 times from baseline up to 12 months: At baseline, day 14, 68, 98, 140, 182, 196, 273 and day 365.
improvement in psychopathology (GAF) | 12 months (At baseline, day 98, 182 and day 365)
  The Social Assessment of Functioning Scale (GAF) also estimates social and professional performance. It takes place at all main measurement times. At baseline, day 98, 182 and day 365.
improvement in psychopathology (BSI-53) | 12 months (At baseline, day 98, 182 and day 365)
  The Brief Symptom Inventory (BSI-53) records the symptoms using 53 items. It takes place at all main measurement times. At baseline, day 98, 182 and day 365.
improvement in psychopathology (CDSS) | 12 months (at baseline, day 14, 68, 98, 140, 182, 196, 273 and day 365)
  The Calgary Depression Scale for Schizophrenia (CDSS) measures suicidality and severity of depressive symptoms. It will be called up 9 times from baseline up to 12 months: At baseline, day 14, 68, 98, 140, 182, 196, 273 and day 365.
improvement in social and occupational functioning (UPSA-B) | 12 months (at baseline, day 98, day 182 and day 365)
  The University of California San Diego Performance-based Skills Assessment (UPSA-B) will be used to assess the day-to-day functioning of patients with schizophrenia in the household, communications, finance, transportation, and leisure activities role play situations. It takes place at all main measurement times. At baseline, day 98, 182 and day 365.
improvement in social and occupational functioning (FROGS) | 12 months (at baseline, day 98, day 182 and day 365)
  Functional Remission of General Schizophrenia (FROGS) is used as a tool to measure changes in functional levels. It takes place at all main measurement times. At baseline, day 98, 182 and day 365.
improvement in social and occupational functioning (PSP) | 12 months (at baseline, day 98, day 182 and day 365)
  The Personal and Social Performance Scale (PSP) is also a tool to measure changes in functional levels. It takes place at all main measurement times. At baseline, day 98, 182 and day 365.
improvement in quality of life | 12 months (at baseline, day 182 and day 365)
  Only at the beginning and end of the intervention, and after one year, is the World Health Organization's Quality of Life Questionnaire (WHOQOL-Bref) used to record quality of life (The WHOQOL Group, 1998).
improvement in body mass index (BMI) | 12 months (at baseline, day 14, 68, 98, 140, 182, 196, 273 and day 365)
  Also, the body height (in meter) and weight (in kg) of the study participants are measured. Thereupon the BMI is calculated from the body weight (kg) divided by the square of the height (m2). The unit of BMI is kg / m2.
change of connectivity analysis (MRI of the brain) | 12 months (at baseline, day 98, day 182 and day 365)
  At four time points, just prior to initiation of V1, V4, V6 after the end of the intervention and at V9 after the follow-up period of 6 months, structural and functional MRI (fMRI) examinations are performed on a 3 Tesla whole-body MR scanner in patients and healthy control subjects (Siemens) made.
  The findings are compared with data from healthy controls and non-diseased first-degree relatives of patients with schizophrenia who have been evaluated in other BMBF-funded studies ("MooDS", "IntegraMent"). In addition, cross-sectional comparisons (TAU + Exercise vs. TAU + BKGT) and progress measurements to characterize treatment effects are planned. The measurements are divided into 2 appointments to reduce the burden on patients and subjects by the measurement time.
change of volumes of brain regions (MRI) | 12 months (at baseline, day 98, day 182 and day 365)
  First, structural measurements (T1 sequence, duration: approx. 5 minutes) and investigations of the fiber connections in the brain by means of diffusion-weighted imaging (DTI, duration: approx. 10 minutes) are carried out.
change of brain function (MRI) | 12 months (at baseline, day 98, day 182 and day 365)
  By means of fMRI, the tasks resting activity, working memory, episodic memory, reward processing, social perspective takeover, emotion processing as well as ability to inhibit are to be investigated with already well pre-examined tasks.
  A function measurement is performed at rest without stimulation (rsMRT), which provides information on the functional networking of different brain regions at rest (duration: approx. 5 minutes). There are also three fMRI surveys that record brain activity during simple psychological tasks. - The ability to inhibit (prefrontal cortex, anterior cingulate gyrus) is examined by means of a so-called flanker task. This is to respond to a specific target stimulus, which is surrounded by either the same (congruent) or by distracting (incongruent) stimuli. - Duration: 11 minutes
improvement of endurance capacity | 12 months (at baseline, day 98, day 182 and day 365)
  As part of the sports medical stress test, the determination of endurance performance in patients and control subjects takes place. For this examination, like in training, finder bike use and measurements of heart rate, lactate concentration and exertion sensation are performed. The ergometry is carried out as a Vita maxima examination, so it ends when the subjects can not or do not want to keep pedaling or when the termination criteria according to Steinacker & Liu (2002) occur. From the examination, various submaximal and maximal parameters can be determined, have the validity for endurance performance and the training intensity can be determined. The examination is carried out under standardized and safe conditions and after a detailed medical history and physical examination to exclude contraindications.
  Activity meters are used to control the physical activity of study participants outside the study intervention.
change of medication and attitude of the study participants to therapy (DAI) | 12 months (at baseline, day 98, day 182 and day 365)
  Also, the attitude of the study participants to therapy and medication is recorded. For this, the Drug Attitude Inventory (DAI) is used. Is takes place at the main measurement times (at baseline, day 98, day 182 and day 365).
change of medication and attitude of the study participants to therapy (SES) | 12 months (at baseline, day 98, day 182 and day 365)
  The Service Engagement Scale (SES), which assesses accessibility, cooperation, help seeking and adherence, is used. It takes place at the main measurement times (at baseline, day 98, day 182 and day 365).
improvement in metabolic parameters | 12 months (at baseline, day 98, day 182 and day 365)
  The laboratory diagnostic measures include a laboratory blood test, with evaluation of blood lipid levels, the C-reactive protein, glycohemoglobin (HBA1c). It takes place at the main measurement times (at baseline, day 98, day 182 and day 365).
urine (testing pregnancy and drug abuse) | baseline
  Examination of the urine at baseline excludes pregnancy and drug abuse.
gene expression | baseline
  Investigation of gene expression takes place at baseline.
change of genome-wide epigenetics | 12 months (at baseline, day 98, day 182 and day 365)
  Investigation of genome-wide epigenetics takes place at the main measurement times (at baseline, day 98, day 182 and day 365).
change of proteomics | 12 months (at baseline, day 98, day 182 and day 365)
  Investigation of proteomics at the main measurement times (at baseline, day 98, day 182 and day 365).
change of BDNF level | 12 months (at baseline, day 98, day 182 and day 365)
  Investigation of BDNF levels at the main measurement times (at baseline, day 98, day 182 and day 365).

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Falkai, Prof. Dr., Principal Investigator — LMU Munich
Locations (1):
- Ludwig-Maximilians-University of Munich, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Schwaiger R, Maurus I, Lembeck M, Papazova I, Greska D, Muenz S, Sykorova E, Thieme CE, Vogel BO, Mohnke S, Huppertz C, Roeh A, Keller-Varady K, Malchow B, Walter H, Wolfarth B, Wolwer W, Henkel K, Hirjak D, Schmitt A, Hasan A, Meyer-Lindenberg A, Falkai P, Roell L. Predictors of adherence to exercise interventions in people with schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2024 Sep;274(6):1265-1276. doi: 10.1007/s00406-024-01789-w. Epub 2024 Mar 29. PMID 38551773
- [Derived] Roell L, Keeser D, Papazov B, Lembeck M, Papazova I, Greska D, Muenz S, Schneider-Axmann T, Sykorova EB, Thieme CE, Vogel BO, Mohnke S, Huppertz C, Roeh A, Keller-Varady K, Malchow B, Stoecklein S, Ertl-Wagner B, Henkel K, Wolfarth B, Tantchik W, Walter H, Hirjak D, Schmitt A, Hasan A, Meyer-Lindenberg A, Falkai P, Maurus I. Effects of Exercise on Structural and Functional Brain Patterns in Schizophrenia-Data From a Multicenter Randomized-Controlled Study. Schizophr Bull. 2024 Jan 1;50(1):145-156. doi: 10.1093/schbul/sbad113. PMID 37597507
- [Derived] Maurus I, Roell L, Keeser D, Papazov B, Papazova I, Lembeck M, Roeh A, Wagner E, Hirjak D, Malchow B, Ertl-Wagner B, Stoecklein S, Hasan A, Schmitt A, Meyer-Lindenberg A, Falkai P. Fitness is positively associated with hippocampal formation subfield volumes in schizophrenia: a multiparametric magnetic resonance imaging study. Transl Psychiatry. 2022 Sep 16;12(1):388. doi: 10.1038/s41398-022-02155-x. PMID 36114184
- [Derived] Roell L, Maurus I, Keeser D, Karali T, Papazov B, Hasan A, Schmitt A, Papazova I, Lembeck M, Hirjak D, Sykorova E, Thieme CE, Muenz S, Seitz V, Greska D, Campana M, Wagner E, Loehrs L, Stoecklein S, Ertl-Wagner B, Poemsl J, Roeh A, Malchow B, Keller-Varady K, Meyer-Lindenberg A, Falkai P. Association between aerobic fitness and the functional connectome in patients with schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2022 Oct;272(7):1253-1272. doi: 10.1007/s00406-022-01411-x. Epub 2022 Apr 30. PMID 35488054
- [Derived] Maurus I, Hasan A, Schmitt A, Roeh A, Keeser D, Malchow B, Schneider-Axmann T, Hellmich M, Schmied S, Lembeck M, Keller-Varady K, Papazova I, Hirjak D, Topor CE, Walter H, Mohnke S, Vogel BO, Wolwer W, Schneider F, Henkel K, Meyer-Lindenberg A, Falkai P. Aerobic endurance training to improve cognition and enhance recovery in schizophrenia: design and methodology of a multicenter randomized controlled trial. Eur Arch Psychiatry Clin Neurosci. 2021 Mar;271(2):315-324. doi: 10.1007/s00406-020-01175-2. Epub 2020 Aug 3. PMID 32748261